CLINICAL TRIAL: NCT06529198
Title: The NEUROGYN-GNS Pivotal Clinical Study to Assess the Safety and Efficacy of the Neurogyn Genital Neuromodulation System, a Genital Nerves Neuromodulation Device Used to Treat Idiopathic Overactive Bladder (iOAB).
Brief Title: NeuroGyn Genital Neuromodulation System for iOAB Treatment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dr. med. Marc Possover (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. med. Marc Possover, PhD MD, Possover International Medical Center AG
Organization: Possover International Medical Center AG (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NeuroGyn AG
Record Dates: First submitted 2024-07-13; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment (Experimental): Patient are undergoing neuromodulatioon
  Interventions: Device: NeuroGyn Genital Neuromodulation System

INTERVENTIONS:
Device: NeuroGyn Genital Neuromodulation System — Genital Neuromodulation

SUMMARY:
The NeuroGyn study is designed to evaluate the safety and effectiveness to the NeuroGyn Genital Neuromodulation System as an aid in the treatment of the symptoms of idiopathic overactive bladder in patients who have failed or could not tolerate more conservative treatments.

DETAILED DESCRIPTION:
not provided

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older (adult and older adult, all sexes)
* Diagnosed (urodynamic testing) with idiopathic overactive bladder (iOAB)
* Symptoms of urinary urgency, frequency, and/or urge incontinence for at least 6 months
* Failed conservative treatments (e.g., lifestyle modifications, medications)
* Willing and capable of providing informed consent
* Capable of participating in all testing associated with this clinical investigation
* Patients have already undergo a successful GNS-test phase with adhesive electrodes (reduction symptoms greater equal or more than 50%)

Exclusion Criteria:

* History of pelvic surgery affecting the pubic bone or genital nerves
* Current urinary tract infection
* Neurological conditions affecting bladder function (neurogenic OAB)
* Pregnancy or planning to become pregnant during the study period
* Contraindications to local anesthesia or surgery
* Female patients with significant prolapse (i.e., prolapse beyond the introitus).
* Patients with primary stress incontinence and primary pelvic pain symptoms.
* Patients with less than 12 months from last intravesical botulinum toxin A therapy
* Patients with mechanical infravesical obstruction and/or Interstitial Cystitis.
* Vulnerable patients with co-morbid conditions should be excluded from this study. These co-morbid conditions include all pathologies of the cardiovascular system (Angina Pectoris, Infarct, Thrombose, Embolie, Hypertonia), pulmonary system (asthma, COPD, chr. Bronchitis), intestinal system (morbus Crohn, diverticulitis..) and any malignant disease. These co-morbid conditions also include neurologic diseases (i.e., stroke, multiple sclerosis, spinal cord injury), sacral dermal pathological conditions, congenital or other anatomical sacral anomalies (e.g. spina bifida, sacral agenesis, trauma sequelae), mobility deficits, medically complicated/uncontrolled diabetes, fecal motility disorders (fecal incontinence/constipation), chronic pelvic pain, history of recurrent urinary tract infections (UTIs), gross hematuria, prior pelvic/vaginal surgeries (incontinence/prolapse surgeries), pelvic cancer (bladder, colon, cervix, uterus, prostate), deeply infiltrating endometriosis of the pelvic plexus, sacral plexus or of the bladder, Reiter´s syndrome, and pelvic radiation.
* Patients suffering from other CNS disorders (mental disorders, severe psychological problems, cerebrovascular accident less than 6 months ago).
* Patients suffering from polydipsia/polyuria are excluded from the study. Similarly, patients suffering from diabetes insipidus (DI) and diabetes mellitus (DM) are also excluded from the study.
* A female with a positive urine pregnancy test
* A female who is breastfeeding
* Allergies again local anesthesia (Lidocain), Tranquillizers and Antibiotics

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — femal and male
Enrollment: 150 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Reduction in Symptoms greater than or equal to 50% | 6 months - 1 year - 2 years follow up
  Overactive Bladder Symptom Score - OABSS
Urodynamic testing | 6 months - 1 year - 2 years
  Noninvasive uroflowmetry, followed by invasive cystometry and a pressure-flow study + concurrent electromyography (EMG) of pelvic floor muscles and urethral pressure profiles

SECONDARY OUTCOMES:
International Consultation on Incontinence Questionnaire | 6 months - 1 year - 2 years
  International Consultation on Incontinence Questionnaire (ICIQ)
The PHQ-9 (Patient Health Questionnaire-9) | 6 months - 1 year - 2 years
  PHQ-9

IPD SHARING:
Plan to Share IPD: No